CLINICAL TRIAL: NCT07225478
Title: Clinical Study to Evaluate the Tooth Whitening Efficacy of a New NextGen In-office Whitening System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2025-09-WHT-MS
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Health Adult Subjects
Keywords: In-Office Whitening; Dental Whitening

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- NextGen In-Office Whitening System (Experimental): Providers will apply NextGen in-office whitening according to detailed instructions included in Appendix XII of the protocol. This includes application of a gingival barrier, followed by application of the whitening gel to the teeth directly for 3 sessions of 15 minutes each. An LED tray will also be worn during these sessions. Afterwards, all gel, barriers and isolation will be removed. Participants will be given a toothbrush and toothbrush for home use, and instructed to brush for 2 minutes twice a day.
  Interventions: Drug: Beaming White; Drug: Fluoride Toothpaste; Device: Soft Manual Toothbrush; Device: CP LED; Device: Gingival Barrier
- Zoom In-Office Whitening System (Active Comparator): Providers will apply Zoom in-office whitening according to the manufacturer's instructions, included in Appendix XII of the protocol. This includes application of a gingival barrier, followed by application of the whitening gel to the teeth directly for 3 sessions of 15 minutes each, and use of the Philips Zoom Whitespeed Lamp. Afterwards, all gel, barriers and isolation will be removed. Participants will be given a toothbrush and toothbrush for home use, and instructed to brush for 2 minutes twice a day.
  Interventions: Combination Product: Philips Zoom Professional Whitening Treatment; Drug: Fluoride Toothpaste; Device: Soft Manual Toothbrush
- Opalescence In-Office Whitening System (Active Comparator): Providers will apply Opalescence in-office whitening according to the manufacturer's instructions, included in Appendix XII of the protocol. This includes application of a gingival barrier, followed by application of the whitening gel to the teeth directly for 3 sessions of 20 minutes each. Afterwards, all gel, barriers and isolation will be removed. Participants will be given a toothbrush and toothbrush for home use, and instructed to brush for 2 minutes twice a day.
  Interventions: Combination Product: Opalescence Boost PF; Drug: Fluoride Toothpaste; Device: Soft Manual Toothbrush

INTERVENTIONS:
Drug: Beaming White — 25%HP gel for in office use only
  Arms: NextGen In-Office Whitening System
Combination Product: Philips Zoom Professional Whitening Treatment — Light-Activated Whitening - Contains 25% HP gel for in-office use only
  Arms: Zoom In-Office Whitening System
Combination Product: Opalescence Boost PF — Contains 40%HP whitening gel for in-office use only
  Arms: Opalescence In-Office Whitening System
Drug: Fluoride Toothpaste — Colgate Cavity Protection Toothpaste
Device: Soft Manual Toothbrush — Colgate Adult Extra Clean soft-bristle toothbrush
Device: CP LED — CP LED 20mA
  Arms: NextGen In-Office Whitening System
Device: Gingival Barrier — Gingival Barrier
  Arms: NextGen In-Office Whitening System

SUMMARY:
The goal of this clinical study is to evaluate how well a new in-office whitening system works to whiten teeth compared to some other commercially available in-office whitening systems.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Male and female subjects aged 18-70 years, inclusive;
* Good general health and good oral health based on the opinion of the study investigator;
* All maxillary natural anterior teeth (teeth #6 through #11) must be present;
* Availability for the duration of the study;
* Minimum average Vita Extended Bleachedguide 3D-Master shade score of 17 ≥ or darker.

Exclusion Criteria:

* Presence of orthodontic appliances and/or any anterior tooth with a prosthetic crown, veneer, or deemed non-vital;
* Obvious signs of periodontal disease, rampant caries, or any condition that the dental examiner considers exclusionary from the study.
* Five or more carious lesions requiring immediate care.
* Concurrent participation in another oral clinical study.
* Self-reported pregnant and/or lactating women.
* History of allergies or sensitivity to tooth whitening products, hydrogen peroxide, personal care consumer products, or their ingredients;
* Restorations on the teeth to be scored which may interfere with scoring procedures.
* Have used professional whitening products within one (1) year and/or had dental prophylaxis (professional dental cleaning) within thirty (30) days prior to the start of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2025-10-31 (Actual); Primary Completion 2025-12-21 (Actual); Study Completion 2025-12-21 (Actual)

PRIMARY OUTCOMES:
Whitening Improvements | Immediately after whitening and 1 week later.
  The primary outcome variable of this study will be tooth shade whitening improvements via the Vita Extended BleachedGuide 3D-Master (29 tabs).

CONTACTS AND LOCATIONS:
Locations (1):
- Consumer Research Consulting, LLC, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: No